CLINICAL TRIAL: NCT02692495
Title: Evaluation of Gastrointestinal and Nutritional Diagnostic Tests as Potential Screening Tools for Metabolic Body Odor and Halitosis
Brief Title: Evaluation of Potential Screening Tools for Metabolic Body Odor and Halitosis
Status: Completed | Type: Observational
Sponsor: Mebo Research, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 200904010001MEBO
Record Dates: First submitted 2016-02-16; First posted 2016-02-26 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: body odor; halitosis; dysbiosis; leaky gut; microbiome; PATM; breath odor
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Body Odor; Halitosis; Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Body odor: individuals self-reporting recurrent episodes of uncontrollable body odor with or without halitosis
- Halitosis: individuals with extra-oral halitosis, not complaining of body odors

SUMMARY:
This study is designed as a retrospective cohort study to evaluate the potential of diagnostic procedures in defining populations of patients self-reporting unexpected and uncontrollable episodes of body odor and/or halitosis. The cohort - generally healthy individuals who had underwent multiple diagnostic tests recommended by their physicians and had not been diagnosed with any known medical condition - expressed their interest in trying gastrointestinal and nutritional diagnostic tests offered by Biolab Medical Unit. Our retrospective analysis will determine if these tests were useful as potential screening tools for metabolic body odor and halitosis.

DETAILED DESCRIPTION:
Many yet uncharacterized medical conditions including inborn and acquired errors of metabolism or skewed microbiome could be responsible for unpredictable and uncontrollable episodes of body odor and halitosis. These conditions have dramatic impact on the quality of life and socioeconomic outcomes of sufferers. Yet clinics and specialized malodor centers do not provide tests for diagnosing malodor other than trimethylaminuria (TMAU). Self-reported odor problems are often dismissed if are not organoleptically evaluated by trained odor judges that are not readily available during malodor flare-ups.

The aim of this study is to analyze effectiveness of existing gastrointestinal and nutritional tests for the assessment and investigation of self-reported malodors.

Diagnostic tests included:

* Gut Permeability Profile. PEG 400 is used as a probe and measured in urine passed for the following 6 hours at 11 different molecular weights to establish the quantity of each absorbed through the gut wall. Extraction and separation of PEG from urine is done by ion exchange chromatography and capillary GLC.
* Gut Fermentation Profile. Blood alcohols - ethanol, methanol, butanol, propanol and short chain fatty acids - are measured by gas-liquid chromatography.
* D-lactate test. D-lactate is measured by centrifugal analysis using the specific enzyme D-lactate dehydrogenase, which does not react with L-lactate
* The urine indicans (Obermeyer) test. Detection of indican in the urine depends upon its decomposition and subsequent oxidation of indoxyl to indigo blue and its absorption into a chloroform layer
* Breath test for small intestinal dysbiosis. Breath hydrogen and methane are measured by gas-liquid chromatography. The patient is given 10 gm of lactulose in 200 ml of water and alveolar air samples are collected every 20 minutes for 3 hours
* Functional B vitamins profile, by measuring the activation of a red cell enzyme that is dependent upon an adequate concentration of a particular vitamin for full activity. The assay relies on normal metabolism of the vitamin to its native form and the presence of other non-vitamin cofactors.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic malodor experienced over a period of several months or years
* willing and able to complete the study
* good general health

Exclusion Criteria:

* elect not to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals reporting idiopathic malodor production
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2013-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Gabashvili, PhD, Principal Investigator — MeBO Research
Locations (1):
- MeBO Research LTD, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data will be made partially available

REFERENCES:
- [Background] Chadwick VS, Phillips SF, Hofmann AF. Measurements of intestinal permeability using low molecular weight polyethylene glycols (PEG 400). I. Chemical analysis and biological properties of PEG 400. Gastroenterology. 1977 Aug;73(2):241-6. PMID 873124
- [Background] Sivakumaran T, Jenkins RT, Walker WH, Goodacre RL. Simplified measurement of polyethylene glycol 400 in urine. Clin Chem. 1982 Dec;28(12):2452-3. No abstract available. PMID 7139937
- [Background] Hunnisett A., Howard J., Davies S. Gut fermentation (or the 'Auto-brewery') Syndrome: A new clinical test with initial observations and discussion of clinical and biochemical implications J.Nutr.Med.1:33-8, 1990
- [Background] Sheedy JR, Wettenhall RE, Scanlon D, Gooley PR, Lewis DP, McGregor N, Stapleton DI, Butt HL, DE Meirleir KL. Increased d-lactic Acid intestinal bacteria in patients with chronic fatigue syndrome. In Vivo. 2009 Jul-Aug;23(4):621-8. PMID 19567398
- [Background] Ludvigsen CW, Thurn JR, Pierpont GL, Eckfeldt JH. Kinetic enzymic assay for D(-)-lactate, with use of a centrifugal analyzer. Clin Chem. 1983 Oct;29(10):1823-5. PMID 6616831
- [Background] Jenq RR. How's your microbiota? Let's check your urine. Blood. 2015 Oct 1;126(14):1641-2. doi: 10.1182/blood-2015-08-661504. PMID 26429966
- [Background] Khoshini R, Dai SC, Lezcano S, Pimentel M. A systematic review of diagnostic tests for small intestinal bacterial overgrowth. Dig Dis Sci. 2008 Jun;53(6):1443-54. doi: 10.1007/s10620-007-0065-1. PMID 17990113
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Mount JN, Heduan E, Herd C, Jupp R, Kearney E, Marsh A. Adaptation of coenzyme stimulation assays for the nutritional assessment of vitamins B1, B2 and B6 using the Cobas Bio centrifugal analyser. Ann Clin Biochem. 1987 Jan;24 ( Pt 1):41-6. doi: 10.1177/000456328702400106. PMID 3827183
- Available data/document: Individual Participant Data Set: 10.17632/8bk6h6bmkr.1 — https://data.mendeley.com/datasets/8bk6h6bmkr/1
- Available data/document: Clinical Study Report — http://www.aurametrix.com/nct02692495
- Available data/document: Preprint: 10.1101/139014 — http://biorxiv.org/content/early/2017/05/19/139014 — Study results

RESULTS

PARTICIPANT FLOW:
Groups:
- Halitosis: individuals with halitosis (bad breath), not complaining of body odors
Period: Overall Study
Arm/Group | Body Odor | Halitosis
Started | 12 | 4
Completed | 12 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Halitosis: individuals with halitosis, not complaining of body odors
- Total: Total of all reporting groups
Arm/Group | Body Odor | Halitosis | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (8.5) | 37.5 (5.9) | 32.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 4 | 16
Duration of condition [Mean (Standard Deviation); unit: years]
  Age at onset of symptoms | 21 (9) | 29 (9) | 23 (9)
  Duration of symptoms | 9 (6) | 9 (5) | 9 (6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Test Results Outside the Normal Range
Description: The investigators would like to evaluate the strength of evidence in diagnostic accuracy of laboratory tests taken by participants (listed in the detailed description of the study), for diagnosing malodor syndromes. Values measured by the laboratory (Biolab Medical Unit) will be compared against the reference range specific to that laboratory.
Time Frame: four years
Measure: Number; unit: participants
Arm/Group | Body Odor | Halitosis
Number analyzed (Participants) | 12 | 4
participants
  Elevated blood ethanol | 6 | 3
  Elevated blood methanol | 0 | 0
  Elevated 1-propanol | 8 | 3
  Elevated 2-propanol | 3 | 3
  Elevated 2-methyl-1-propanol | 6 | 2
  Elevated 2-methyl-2-propanol | 0 | 1
  Elevated 1-butanol | 1 | 0
  Elevated 2-butanol | 2 | 0
  Elevated 2-methyl-1-butanol | 6 | 1
  Elevated 2-methyl-2-butanol | 0 | 0
  Elevated 2-ethyl-1-butanol | 0 | 1
  Elevated 2,3-butylene glycol | 4 | 0
  Increased blood acetate | 0 | 1
  Decreased blood acetate | 4 | 0
  Decreased blood propionate | 4 | 0
  Decreased blood butyrate | 5 | 0
  Blood Succinate out of range | 0 | 0
  Blood Valerate out of range | 0 | 0
  Increased gut permeability | 9 | 0
  Decreased gut permeability | 0 | 2
  increased blood D-lactate | 3 | 0
  increased urine Indicans | 5 | 1

2. Secondary Outcome: Discriminative Biomarkers in the Subgroups of Malodor
Description: The investigators have comprehensively analyzed diagnostic ability of tests taken by participants to correlate with their symptoms using several statistical techniques known to bring out strong patterns in a dataset. Principal component analysis (PCA) allowed to clearly separate data into two clusters ("Sour" and "Sweet") shown below along with the "Lactic" subgroup from the "Sour" group.
Time Frame: three years
Measure: Mean (Standard Deviation); unit: umol/L
Groups:
- "Sour" Group: Self-reported predominant odors included "fishy", "ammonia", sour acetone (body odor associated with alcoholism), fecal-diarrheal, and generic "fecal odor"
- "Sweet" Group: Self-reported odors mostly identified as gas, benzene, "burning","sulfur", "rotten vegetables", "rotten eggs", cheesy/sweaty and sulfury fecal, sewage, "burning", and elusive odors that could not be smelled by the sufferer including "PATM" condition (odors could not be named, but people near the sufferer exhibited increased displeasure, coughing, sneezing, and rubbing their noses).
- "Lactic" Subgroup: "Garbage" odor identified as one of the most common types of odor (subgroup of the "Sour" cluster)
Arm/Group | "Sour" Group | "Sweet" Group | "Lactic" Subgroup
Number analyzed (Participants) | 7 | 7 | 2
umol/L
  D-lactate | 7 (5) | 29 (39) | 330 (245)
  2- butanol | 1.3 (0.8) | 0.9 (0.7) | 3.2 (1.2)
  Butyrate | 5 (6) | 11 (3) | 6 (6)
  2,3-butylene glycol | 2.6 (1.4) | 1.6 (1.5) | 6.0 (0.0)
  Acetate | 60.6 (16.9) | 68.7 (22.5) | 55.5 (37.5)
Statistical Analysis 1: Comparison: "Sour" Group vs "Sweet" Group vs "Lactic" Subgroup; Test type: Other; p < 0.01, t-test, 2 sided

3. Secondary Outcome: Number of Test Results Outside the Normal Range in Different Subgroups of Malodor
Description: Disciminative biomarkers for groups of malodor discovered using PCA, compared to control group
Time Frame: Three years
Measure: Count of Participants; unit: Participants
Groups:
- "Lactic" Subgroup: "Garbage" odor identified as one of the most common types of odor
Arm/Group | "Sour" Group | "Sweet" Group | "Lactic" Subgroup
Number analyzed (Participants) | 7 | 7 | 2
Participants
  Ethanol, blood | 0 | 7 | 1
  Indicans, urine | 1 | 4 | 1
  B2 vitamin, blood (EGFR activation) | 1 | 5 | 0
  D lactate, plasma | 0 | 0 | 2

4. Secondary Outcome: Average Daily Added Sugar Intake Inferred From Self-reported Dietary Data in the Subgroups of Malodor
Description: The measurement of dietary intake of selected nutrients from self-reported food intakes and diet history questionnaires. Correlation of symptoms with added sugar in the diet were noted independently on the source of malodor.
Time Frame: Three years
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | "Sour" Group | "Sweet" Group | "Lactic" Subgroup
Number analyzed (Participants) | 7 | 7 | 2
grams per day | 5 (5) | 25 (10) | 20 (10)

ADVERSE EVENTS:
Time Frame: All participants were followed up by email for at least one week after discussing their test results.
Description: Adverse effects were defined as any events, expected or not, that affected participant well being, regardless of whether there was a causal relationship with the diagnostic testing and discussion of the results.
  Serious adverse events were defined as those that prevented a participant from performing normal activities and required treatment.
Groups:
- Halitosis: individuals self-reporting breath malodors but not body odors
Arm/Group | Body Odor | Halitosis
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 0/12 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes